CLINICAL TRIAL: NCT04963699
Title: The Study of N-terminal Pro-brain Natriuretic Peptide Combined With High-sensitivity Troponin T in Evaluating the Prognosis of Sepsis
Brief Title: The Study of NT-proBNP Combined With HS-cTnT in Evaluating the Prognosis of Sepsis
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0317
Record Dates: First submitted 2021-06-09; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2016-06

CONDITIONS: Sepsis
Keywords: N-terminal pro-brain natriuretic peptide; High-sensitivity troponin T
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
To study the clinical value of combined detection of plasma N-terminal pro-brain natriuretic peptide (NT-proBNP) and high-sensitivity troponin T (hs-cTnT) in assessing the prognosis of patients with sepsis. Methods Seventy-three patients with sepsis who were diagnosed and treated in our hospital from June 2016 to March 2021 were divided into general sepsis group and severe sepsis group. According to different outcomes, they were divided into survival Group and death group, to explore the relationship between plasma NT-proBNP, hs-cTnT levels and APACHEⅡ score and the value of prognostic evaluation of sepsis.

DETAILED DESCRIPTION:
1.1 Information The 73 patients with sepsis who were diagnosed and treated in our hospital from June 2016 to March 2021 were selected as the research objects. All of them had clear infections through clinical examination; there were no acute coronary syndromes, no immunodeficiency diseases, and no immunodeficiency diseases in the past month. No tumors, etc.; no pulmonary embolism and aortic dissection; no valvular heart disease, cardiomyopathy, myocarditis, etc.; no pregnant women and lactating women; no congenital heart, liver, kidney and other organ diseases. The diagnostic criteria of sepsis refer to the "Guidelines for the Emergency Treatment of Sepsis/Septic Shock in China (2018)" [5]. The patients were divided into general sepsis group (30 cases) and severe sepsis group (43 cases) according to the severity of their illness. The severe sepsis group included severe sepsis (35 cases) and septic shock (8 cases). , Select the population (40 cases) in our hospital for physical examination during the same period as the healthy control group.

1.2 Method 1.2.1 Testing equipment: All patients with sepsis will take 3ml of cubital venous blood when they are admitted to the hospital and place them in a green-head tube containing lithium heparin anticoagulant produced by BD in the United States. After centrifugation at 3000 r/min for 10 minutes, they will be tested immediately; health In the control group, 3ml of cubital venous blood was drawn on an empty stomach in the morning of the physical examination, placed in a lithium heparin anticoagulation tube, centrifuged at 3000 r/min for 10 minutes, and the test was completed within 2 hours. Choose Roche cobas e 601 electrochemiluminescence immunoassay analyzer to detect blood NT-pro BNP and hs-cTnT. Mindray BC 6900 blood cell analyzer detects white blood cell count, Beckman Coulter 5831 automatic biochemical analyzer detects C-reactive protein; all operations are performed in strict accordance with the reagent instructions.

1.2.2 Observation indicators Patients with sepsis undergo acute physiological and chronic health assessment (APACHE II score) within 24 hours after diagnosis.

1.3 Statistical processing SPSS 23.0 software was used for data statistical analysis, measurement data application (x ± s) description, non-parametric test Mann-Whitney U test was used for comparison between groups; plasma NT-proBNP and hs-cTnT were analyzed by rank correlation analysis The correlation between the level and the APACHEⅡ score was analyzed, and the Spearman rank correlation coefficient was used to describe the correlation.

ELIGIBILITY:
Inclusion Criteria:

* All have clear infection through clinical examination; no acute coronary syndrome, no immunodeficiency, no tumor, etc. in the past 1 month; no pulmonary embolism or aortic dissection; no valvular heart disease, cardiomyopathy, myocarditis, etc.; no pregnant women And lactating women; no congenital heart, liver, kidney and other organ diseases.

Exclusion Criteria:

* Acute coronary syndrome, immunodeficiency, tumor, etc. in the past month; pulmonary embolism and aortic dissection; valvular heart disease, cardiomyopathy, myocarditis, etc.; pregnant and lactating women; congenital Heart, liver, kidney and other organ diseases

Ages: 16 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with sepsis who were diagnosed and treated in our hospital from June 2016 to March 2021
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
NT-proBNP | 2016.06.01-----2021.03.30
  NT-proBNP is used as an aid to diagnose and monitor mild cardiac dysfunction in individuals suspected of having congestive heart failure. Compared with BNP, NT-proBNP has a longer half-life, better stability, and higher plasma concentration. , Has superiority in predicting myocardial function. Studies have found that NT-proBNP can be used as an important indicator for the prognosis of sepsis with impaired cardiac function and sepsis.The higher the plasma concentration of NT-proBNP, the worse the prognosis.
hs-cTnT | 2016.06.01-----2021.03.30
  hs-cTnT is an independent prognostic marker that can predict the short-term, mid-term and even long-term outcomes of patients with acute coronary syndrome (ACS). Patients with sepsis often have different degrees of damage to myocardial cells, and their plasma hs-cTnT concentration will also increase to different degrees.
APACHEⅡ score | 2016.06.01-----2021.03.30
  During the diagnosis and treatment of sepsis, the APACHE II score can be used to assess the severity of the patient's condition, and is also of important value for the patient's prognostic effect. The higher the score, the more severe the condition.

CONTACTS AND LOCATIONS:
Overall Officials: yang xufeng, MS, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Roche 601 Biochemical Immunoassay Instrument, Hangzhou, Zhejiang, China